CLINICAL TRIAL: NCT01481662
Title: Epidemiological, Clinical and Etiological Features of SUSAC's Syndrome (RETINOCOCHLEOCEREBRAL Vasculopathy)
Brief Title: Epidemiological, Clinical and Etiological Features of SUSAC's Syndrome
Acronym: CARESS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P081261; AOM09039 (Other: french ministery)
Record Dates: First submitted 2011-11-22; First posted 2011-11-29 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-06

CONDITIONS: SUSAC's Syndrome; Encephalopathy; Hearing Loss; Retinal Artery Branch Occlusions
Keywords: SUSAC's Syndrome; encephalopathy; hearing loss; retinal artery branch occlusions; Diffusion tensor MRI
MeSH Terms: conditions — Susac Syndrome; Brain Diseases; Hearing Loss | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — * serum sample
  * cerebrospinal fluid sample
  * DNA sample
  * RNA sample
  * Peripheral Blood Mononuclear Cell sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- retrospective: cases retrospectively reported the last 20 years
- Prospective: Diffusion tensor magnetic resonance imaging of the brain:
  new cases prospectively reported
  Interventions: Device: Diffusion tensor magnetic resonance imaging of the brain

INTERVENTIONS:
Device: Diffusion tensor magnetic resonance imaging of the brain — Diffusion tensor magnetic resonance imaging of the brain will be obtained to more carefully study the cerebral microvasculopathy of the disease.
  Other Names: Diffusion tensor MRI
  Groups: Prospective

SUMMARY:
SUSAC's Syndrome (SS) is characterized by the clinical triad of encephalopathy, hearing loss, and retinal artery branch occlusions. Since the first description of SS in 1979, hundreds of patients with SS, mostly young women, have been reported. However, comprehensive epidemiological, clinical and etiological features of SS have never been specifically addressed so far.

The objective of this study is to characterize the epidemiological, clinical, and etiological features of SUSAC's Syndrome. In this aim, the investigators will constitute a national clinical-based cohort including all SS cases retrospectively reported in France since the last 20 years and all new cases prospectively observed. French Society of Neurology, Ophthalmology and Internal Medicine will be asked to collaborate. Every case will be reviewed by an expert comity of internists, neurologists and neuroradiologists to validate the diagnosis. The exhaustive and systematic analysis of each case will help to better define different aspects of the disease such as the incidence and prevalence, the clinical presentation, the diagnostic modalities and the impact of treatments. Diffusion tensor magnetic resonance imaging of the brain will be obtained to more carefully study the cerebral microvasculopathy of the disease. Serum, cerebrospinal fluid, and DNA samples from each patient will also be collected to study potential autoimmune, thrombotic and infectious markers.

DETAILED DESCRIPTION:
SUSAC's Syndrome (SS) is characterized by the clinical triad of encephalopathy, hearing loss, and retinal artery branch occlusions. Since the first description of SS in 1979, hundreds of patients with SS, mostly young women, have been reported. However, comprehensive epidemiological, clinical and etiological features of SS have never been specifically addressed so far.

The diagnosis of SS is difficult because its characteristic signs often do not occur simultaneously or may be too subtle for the patient to notice. Neurological features of SS may occur several months prior to other symptoms. The retinal artery branch occlusion, by occurring in the peripheral portion of the retina, may remain asymptomatic. Sensorineural hearing loss may also be asymptomatic and disclosed only by audiogram. Besides mild pleocytosis in cerebrospinal fluid, all performed biological tests are virtually negative. No infectious agent, consistent autoimmune marker, or coagulopathy has been disclosed. Changes seen on brain MRI are well characterized although not specific. The only site from which biopsy material is available for pathological analysis is the brain. The most common finding in brain biopsies is the presence of microinfarcts but brain biopsy is not currently performed.

Although the treatment of SS has not been studied in controlled trials, most patients have a good response to treatment with glucocorticoids, with the addition of anti-thrombotic therapy and, for cases in which the disease is refractory to steroids, intravenous immune globulin or cyclophosphamide. The clinical course is characterized by recurrent attacks involving 1 or more components of the triad that characterize the active phase of the disease. Remission usually occurs after the active phase but some patients show residual mild to moderate dementia or gait disturbance, and impaired hearing and vision.

SUSAC's Syndrome is a vasculopathy causing small infarcts in the cochlea, retina and brain. Proposed explanations include a hypercoagulable state, vasospasm, and vasculitis, none of which are supported by laboratory results or findings on brain biopsies. The unique distribution of arteriolar disease affecting the brain, the retina, and the cochlea suggests selective vulnerability of these three structures. The brain, retina, and cochlea all have a blood-tissue barrier, and the endothelium in these sites shares a common embryologic origin and unique structural and antigenic characteristics. It has therefore been proposed that SS is an autoimmune disease in which the endothelium is the primary target, and damage to the endothelium triggers arteriolar occlusion and microinfarcts. However, the pathogenesis remains unknown.

The objective of this study is to characterize the epidemiological, clinical, and etiological features of SUSAC's Syndrome. In this aim, we will constitute a national clinical-based cohort including all SS cases retrospectively reported in France since the last 20 years and all new cases prospectively observed. French Society of Neurology, Ophthalmology and Internal Medicine will be asked to collaborate. Every case will be reviewed by an expert comity of internists, neurologists and neuroradiologists to validate the diagnosis. The exhaustive and systematic analysis of each case will help to better define different aspects of the disease such as the incidence and prevalence, the clinical presentation, the diagnostic modalities and the impact of treatments. Diffusion tensor magnetic resonance imaging of the brain will be obtained to more carefully study the cerebral microvasculopathy of the disease. Serum, cerebrospinal fluid, DNA samples from each patient will also be collected to study potential autoimmune, thrombotic and infectious markers.

Because SUSAC's syndrome is a rare disease, we expect to include one hundred patients in this cohort. The constitution of the cohort and the collection of the samples will last for 2 years and half.

The conclusion of the study, based on statistical analysis done once all patients will be included in the cohort, should allow new recommendations in the diagnosis strategy and give new understandings of the therapeutic management of the disease. The result of this study may also give rise to hypothesis for an interventional study.

It's important to underline that this study must be considered as an interventional study.

Indeed, in this study the patients have a specific MRI, the acquisition of the sequences is with diffusion tensor. While in common practice the patients have only classical MRI without this specific sequences which is the routinely technique used.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age older than 18
* Two clinical features of the triad present: encephalopathy, sensorineural hearing loss assessed by audiogram, retinal artery occlusion assessed by fundoscopy or fluorescein retinal angiography.
* Written informed consent provided. In case of subjects unable to give a written informed consent because of encephalopathy associated with the disease, a written statement of non-opposition should be signed by a relative. This non-opposition statement should be then confirmed by the subject as soon as possible.
* Realization of a medical examination beforehand

EXCLUSION CRITERIA:

* Alternative diagnosis: multiple sclerosis, mitochondriopathy, Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leukoencephalopathy (CADASIL), primary brain tumor, Lyme disease.
* In case of associated disease (autoimmune disease, tumor, metabolical disease,…), inclusion will need further analysis by the expert comity.
* Not membership in a national insurance scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SUSAC's Syndrome (SS) is characterized by the clinical triad of encephalopathy, hearing loss, and retinal artery branch occlusions. Hundreds of patients with SS, mostly young women, have been reported.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
To characterize the epidemiological, clinical, and etiological of SUSAC's Syndrome | 1 year
  To characterize the epidemiological, clinical, and etiological of SUSAC's Syndrome

SECONDARY OUTCOMES:
diffusion MRI | 12 months
  diffusion MRI results
serum sample | day 1
  all samples from each patient will be collected to study potential autoimmune, thrombotic and infectious markers
cerebrospinal fluid sample | day 1
  all samples from each patient will be collected to study potential autoimmune, thrombotic and infectious markers
DNA sample | day 1
  all samples from each patient will be collected to study potential autoimmune, thrombotic and infectious markers
RNA sample | day 1
  all samples from each patient will be collected to study potential autoimmune, thrombotic and infectious markers
To characterize the epidemiological, clinical, and etiological of SUSAC's Syndrome | 5 years
  To characterize the epidemiological, clinical, and etiological of SUSAC's Syndrome
Peripheral Blood Mononuclear Cell | 1 day
  all samples from each patient will be collected to study potential autoimmune, thrombotic and infectious markers

CONTACTS AND LOCATIONS:
Overall Officials: Thomas PAPO, Pr, Principal Investigator — APHP
Locations (1):
- Hospital BICHAT, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gaudemer A, Henry-Feugeas MC, Peyre M, Kachaner A, Klein I, Khalil A, Papo T, Sacre K. Brain microstructural damage through serial diffusion tensor imaging and outcomes in Susac syndrome: A prospective cohort study. Eur J Neurol. 2025 Jan;32(1):e70002. doi: 10.1111/ene.70002. PMID 39686647
- [Derived] Kachaner A, Mageau A, Goulenok T, Francois C, Delory N, Chauveheid MP, Laouenan C, Doan S, Halimi C, Klein I, Papo T, Sacre K; French Susac Study Group. Immunosuppressive agents or intravenous immunoglobulin in addition to glucocorticoids in the treatment of Susac syndrome: a French national cohort study. Lancet Rheumatol. 2025 Jan;7(1):e15-e20. doi: 10.1016/S2665-9913(24)00220-0. Epub 2024 Sep 18. PMID 39305913
- [Derived] Scheifer C, Henry Feugeas MC, Roriz M, Cohen Aubart F, Doan S, Jouvent E, Klein I, Machado C, Rouzaud D, Papo T, Sacre K; French Susac Study Group. Brain magnetic resonance imaging lesion load at diagnosis, severity at onset and outcomes in Susac syndrome: A prospective cohort study. Eur J Neurol. 2022 Jan;29(1):121-129. doi: 10.1111/ene.15062. Epub 2021 Aug 23. PMID 34382290
- [Derived] David C, Papo T, Ba I, Ollivier E, Boileau C, Dieude P, Keren B, Kannengiesser C, Sacre K. Hunting for the genetic basis of Susac syndrome. Eur J Neurol. 2021 Jul;28(7):e57-e59. doi: 10.1111/ene.14836. Epub 2021 Apr 7. No abstract available. PMID 33773011
- [Derived] Machado S, Jouvent E, Klein I, De Guio F, Machado C, Cohen-Aubart F, Sacre K, Papo T. Cognitive dysfunction and brain atrophy in Susac syndrome. J Neurol. 2020 Apr;267(4):994-1003. doi: 10.1007/s00415-019-09664-8. Epub 2019 Dec 11. PMID 31828475